CLINICAL TRIAL: NCT00148616
Title: Memantine add-on to Risperidon for Treatment of Negative Symptoms and Cognitive Dysfunction in Patients With Chronic Schizophrenia: Results of a Proof of Concept Study
Brief Title: Memantine for the Treatment of Cognitive Dysfunction and Negative Symptoms in Patients With Chronic Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: M. Schaefer, MD (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, M. Schaefer, MD, Professor of Psychiatry, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIND 2; 02T-247 (SMRI)
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Chronic Schizophrenia
Keywords: Memantine; Negative Syndrome; Schizophrenia; Cognitive impairment
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine plus Risperidone (Active Comparator): 24 weeks memantine add on treatment to risperidone
  Interventions: Drug: Memantine
- Placebo plus Risperidone (Placebo Comparator): 24 weeks placebo add on treatment to risperidone
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Memantine — Daily dosage of 20 mg Memantine add-on to Risperidone vs. Placebo add-on to Risperidone
  Other Names: Akatinol
  Arms: Memantine plus Risperidone
Drug: Placebos — Daily dosage of 20 mg Placebo add-on to Risperidone vs. Memantine add-on to Risperidone
  Other Names: Placebo
  Arms: Placebo plus Risperidone

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 24 weeks memantine add-on treatment to risperidone for the treatment of negative symptomatology and cognitive impairment in patients with chronic schizophrenia.

DETAILED DESCRIPTION:
This study examines the efficacy and safety of 24 weeks memantine add-on treatment to risperidone for the treatment of negative symptomatology and cognitive impairment in patients with chronic schizophrenia. The trail was double-blind, prospective, randomized, placebo-controlled, parallel-group and consisting of a 'placebo-run-in' period, treatment, and follow-up periods. Study personnel and participants were blinded to group assignment. In the 'run-in' period, patients received Lorazepam for the treatment of anxiety and tension states for two weeks before starting antipsychotic therapy. After the 'run-in' period treatment, patients began receiving antipsychotic therapy with Risperidon with continuous concomitant administration of a 24 weeks Memantine, 20 mg/d, or placebo. Adherence was assessed at each clinic visit by pill count. In cases of anxiety and tension states, an experienced psychiatrist decided whether patients should receive Lorazepam, 5 mg/d, as rescue medication in addition to the study medication (Memantine or placebo), to which the patients remained blinded. In cases of pseudo parkinsonism patients were allowed to receive Biperiden, up to 8 mg/d, and for the treatment of patients suffering from sleep disorders Zopiclon (15 mg/d) was allowed. The consumption of alcohol and drugs were not allowed during the trial. In both study parts, psychiatric assessments were performed at baseline as well as after 2; 4; 6; 12 and 24 weeks after treatment (that is, during the follow-up period). The neuropsychological examination was performed at baseline, and after 6 and 24 weeks. Psychiatric changes, adverse events, laboratory values, dose adjustments of the antipsychotic therapy, and possible pharmacologic adverse effects were systematically monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (DSM-IV)
* Age 18 to 40
* Stable negative syndrome (PANSS negative score > 20)
* At least one previous schizophrenic episode
* Informed consent
* Subjects must be considered by the investigator to be compliant with investigations and appointments
* Subjects must have an educational level and a degree of understanding such that they can meaningfully communicate with the investigator

Exclusion Criteria:

* Axis I disorder other than schizophrenia within 12 months, e.g. schizoaffective disorder
* Severe positive symptomatology (PANNS positive score > PANNS negative score)
* Dependency on alcohol or addictive drugs within 6 months of the baseline evaluation
* Contraindication of risperidone
* Significant neurological, cardiovascular, hepatic, renal, metabolic, or other medical diseases or any clinically relevant abnormalities in laboratory tests

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2004-04; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in PANSS negative subscore between memantine and placebo treatment | during trial

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schaefer, MD, Principal Investigator — Charite Campus Mitte; Dept. of Psychiatry and Psychotherapy and Department of Psychiatry, Kliniken Essen-Mitte, Essen
Locations (1):
- Charité Universitaetsmedizin Berlin; Campus Charité Mitte; Dept. for Psychiatry and Psychotherapy, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schaefer M, Sarkar S, Theophil I, Leopold K, Heinz A, Gallinat J. Acute and Long-term Memantine Add-on Treatment to Risperidone Improves Cognitive Dysfunction in Patients with Acute and Chronic Schizophrenia. Pharmacopsychiatry. 2020 Jan;53(1):21-29. doi: 10.1055/a-0970-9310. Epub 2019 Aug 7. PMID 31390660